CLINICAL TRIAL: NCT03734393
Title: HOPE in Action Prospective Multicenter, Clinical Trial of HIV+ Deceased Donor Liver Transplants for HIV+ Recipients
Brief Title: HOPE in Action Trial of HIV+ Deceased Donor Liver Transplants for HIV+ Recipients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00194582; U01AI138897 (NIH)
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIV D+/R+ (Experimental): HIV-infected individuals that accept an organ from an HIV-infected deceased donor - enrollment 40
  Interventions: Other: HIVD+/R+
- HIVD-/R+ (No Intervention): HIV-infected individuals that accept an organ from an HIV-uninfected deceased donor and are randomized to participate in the full study arm, which includes research sample collection -enrollment 40
- HIVD-/R+ (observational) (No Intervention): HIV-infected individuals that accept an organ from an HIV-uninfected deceased donor and randomized to observational group with limited data collection - enrollment 120

INTERVENTIONS:
Other: HIVD+/R+ — Liver from an HIV-infected deceased donor
  Arms: HIV D+/R+

SUMMARY:
The primary objective of this study is to determine if an HIV-infected donor liver (HIVD+) transplant is safe with regards to major transplant-related and HIV-related complications

DETAILED DESCRIPTION:
This study will evaluate if receiving a liver transplant from an HIV-infected deceased liver donor is safe with regards to survival and major transplant-related and HIV-related complications compared to receiving a liver from an HIV-uninfected deceased liver donor (HIVD-). Those participants who have accepted an HIVD- organ will be randomized to be followed in the full study or followed in the nested observational group

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the standard criteria for liver transplant at the local center.
* Participants being listed for a simultaneous liver kidney (SLK) are eligible if participants meet the standard criteria for both organs.
* Participant is able to understand and provide informed consent.
* Participant meets with an independent advocate per the HIV Organ Policy Equity (HOPE) Act Safeguards and Research Criteria.
* Documented HIV infection (by any licensed assay or documented history of detectable HIV-1 RNA).*
* Participant is ≥ 18 years old.
* Opportunistic complications: prior history of certain opportunistic infections is not an exclusion if the participant has received appropriate therapy and has no evidence of active disease. Medical record documentation should be provided whenever possible.
* CD4+ T-cell count: ≥ 100/µL within 16 weeks prior to transplant if no history of AIDS-defining infection; or ≥ 200 μL if history of opportunistic infection is present.
* HIV-1 RNA is below 50 RNA/mL.* Viral blips between 50-400 copies will be allowed as long as there are not consecutive measurements > 200 copies/mL. *Organ recipients who are unable to tolerate anti-retroviral therapy (ART) due to organ.

failure or recently started ART may be eligible despite a detectable viral load if safe and effective ART to be used by the recipient after transplantation is described.

* Participant must have or be willing to start seeing a primary medical care provider with expertise in HIV management.
* Participant is willing to comply with all medications related to participant's transplant and HIV management.
* For participants with a history of aspergillus colonization or disease, no current clinical evidence of active disease.
* Agreement to use contraception.
* Participant is not suffering from significant wasting (e.g. body mass index < 21) thought to be related to HIV disease.

Exclusion Criteria:

* Participant has a history of progressive multifocal leukoencephalopathy (PML), or primary central nervous system (CNS) lymphoma.*
* Participant is pregnant or breastfeeding. (Note: Participants who become pregnant post-transplant will continue to be followed in the study and will be managed per local site practice. Women that become pregnant should not breastfeed.)
* Past or current medical problems or findings from medical history, physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to first death or graft failure or serious adverse event (SAE) or HIV breakthrough or opportunistic infection as a composite measure | From date of transplant through administrative censorship at study completion, up to 4 years
  Time (in days) to first of any of the following events: death or graft failure or SAE or HIV breakthrough or opportunistic infection

SECONDARY OUTCOMES:
Time to Pre-transplant mortality | From date of enrollment to date of transplant or death of any cause, whichever comes first, assessed up to 4 years
  Time (in days) to mortality while enrolled before transplant (survival framework)
Graft Failure as assessed by Time to first occurrence of mortality or re-transplant or return to maintenance dialysis | From date of transplant through administrative censorship at study completion, up to 4 years
  Time (in days) to mortality or re-transplant or return to maintenance dialysis (survival framework)
1-year acute liver rejection | From date of transplant to end of year 1
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2016 comprehensive Update for antibody mediated rejection and Banff 1997 criteria for acute cellular rejection, liver.
2-year acute liver rejection | From date of transplant to end of year 2
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2016 comprehensive Update for antibody mediated rejection and Banff 1997 criteria for acute cellular rejection, liver.
3-year acute liver rejection | From date of transplant to end of year 3
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2016 comprehensive Update for antibody mediated rejection and Banff 1997 criteria for acute cellular rejection, liver.
Number of graft rejections in liver transplant | From date of transplant to end of year 3
  Cumulative incidence of acute rejection (survival framework) as measured by biopsy using Banff 2016 comprehensive Update for antibody mediated rejection and Banff 1997 criteria for acute cellular rejection, liver.
6-month acute kidney rejection in simultaneous liver/kidney transplant recipients | From date of transplant to 6 months post transplant
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2015 criteria: Borderline changes: 'Suspicious' for acute T-cell mediated rejection.This category is used when no intimal arteritis is present, but there are foci of mild tubulitis (t1, t2, or t3) with minor interstitial infiltration (i0 or i1) or interstitial infiltration (i2, i3) with mild (t1) tubulitis. Acute T-cell mediated rejection:Grade from IA defined as cases with significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of moderate tubulitis (t2) to III defined as cases with 'transmural' arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3)
1-year acute kidney rejection in simultaneous liver/kidney transplant recipients only | From date of transplant to end of year 1
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2015 criteria: Borderline changes: 'Suspicious' for acute T-cell mediated rejection.This category is used when no intimal arteritis is present, but there are foci of mild tubulitis (t1, t2, or t3) with minor interstitial infiltration (i0 or i1) or interstitial infiltration (i2, i3) with mild (t1) tubulitis. Acute T-cell mediated rejection:Grade from IA defined as cases with significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of moderate tubulitis (t2) to III defined as cases with 'transmural' arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3)
Number of Non-alcoholic fatty liver (NAFL) | From date of transplant through end of follow-up, up to 3 years
  Cumulative incidence of NAFL as measured by biopsy and transient elastography with controlled attenuation parameter for steatosis
Number of steatohepatitis (NASH) | From date of transplant through end of follow-up, up to 3 years
  Cumulative incidence of NASH as measured by biopsy and transient elastography with controlled attenuation parameter for steatosis
Trajectory of recipient Cluster of Differentiation (CD4) count over time | From date of transplant through end of follow up, up to 4 years
  Analysis of repeated measures of CD4 (cells/mm3) count (longitudinal model)
Trajectory of recipient plasma HIV RNA over time | From date of transplant through end of follow-up, up to 4 years
  Analysis of repeated measures of plasma HIV RNA (copies/mL) longitudinal model
Graft function as assessed by Fibrosis-4 index | 1 years post-transplant
  Mean calculated fibrosis-4 index (Age (years) + AST/platelet count (109/L) x √ALT) Fibrosis 4 index estimates the amount of scar or fibrosis in the liver without requiring a biopsy. Using a lower cutoff value of 1.45, a Fibrosis-4 score <1.45 had a negative predictive value of 90% for advanced fibrosis. In contrast, a Fibrosis-4 >3.25 would have a 97% specificity and a positive predictive value of 65% for advanced fibrosis. In the patient cohort in which this formula was first validated, at least 70% patients had values <1.45 or >3.25.
Graft function as assessed by Fibrosis-4 index | 2 years post-transplant
  Mean calculated fibrosis-4 index (Age (years) + AST/platelet count (109/L) x √ALT) Fibrosis 4 index estimates the amount of scar or fibrosis in the liver without requiring a biopsy. Using a lower cutoff value of 1.45, a Fibrosis-4 score <1.45 had a negative predictive value of 90% for advanced fibrosis. In contrast, a Fibrosis-4 >3.25 would have a 97% specificity and a positive predictive value of 65% for advanced fibrosis. In the patient cohort in which this formula was first validated, at least 70% patients had values <1.45 or >3.25.
Graft function as assessed by Fibrosis-4 index | 3 years post-transplant
  Mean calculated fibrosis-4 index (Age (years) + AST/platelet count (109/L) x √ALT) Fibrosis 4 index estimates the amount of scar or fibrosis in the liver without requiring a biopsy. Using a lower cutoff value of 1.45, a Fibrosis-4 score <1.45 had a negative predictive value of 90% for advanced fibrosis. In contrast, a Fibrosis-4 >3.25 would have a 97% specificity and a positive predictive value of 65% for advanced fibrosis. In the patient cohort in which this formula was first validated, at least 70% patients had values <1.45 or >3.25.
Graft function as assessed by Fibrosis-4 index | 4 years post-transplant
  Mean calculated fibrosis-4 index (Age (years) + AST/platelet count (109/L) x √ALT) Fibrosis 4 index estimates the amount of scar or fibrosis in the liver without requiring a biopsy. Using a lower cutoff value of 1.45, a Fibrosis-4 score <1.45 had a negative predictive value of 90% for advanced fibrosis. In contrast, a Fibrosis-4 >3.25 would have a 97% specificity and a positive predictive value of 65% for advanced fibrosis. In the patient cohort in which this formula was first validated, at least 70% patients had values <1.45 or >3.25.
Graft function as assessed by incidence of fibrosis | From date of transplant through end of follow-up, up to 3 years
  Cumulative incidence of advanced fibrosis (stage F3 or greater as defined by metavir fibrosis score) as measured on biopsy. The fibrosis score is assessed on a five point scale (F0 = no fibrosis, F1 = portal fibrosis without septa, F2 = few septa, F3 = numerous septa without cirrhosis, F4 = cirrhosis).
Graft function as assessed by liver stiffness | 1 year post-transplant
  Mean calculated liver stiffness by transient elastography (kPA)
Graft function as assessed by liver stiffness | 2 years post-transplant
  Mean calculated liver stiffness by transient elastography (kPA)
Graft function as assessed by liver stiffness | 3 years post-transplant
  Mean calculated liver stiffness by transient elastography (kPA)
Average graft function as assessed by aspartate aminotransferase (AST) | 1 year post-transplant
  Mean calculated AST (U/L)
Average graft function as assessed by AST | 2 years post-transplant
  Mean calculated AST (U/L)
Average graft function as assessed by AST | 3 years post-transplant
  Mean calculated AST (U/L)
Average graft function as assessed by AST | 4 years post-transplant
  Mean calculated AST (U/L)
Average graft function as assessed by alanine aminotransferase (ALT) | 1 year post-transplant
  Mean calculated ALT (U/L)
Average graft function as assessed by ALT | 2 years post-transplant
  Mean calculated ALT (U/L)
Average Graft function as assessed by ALT | 3 years post-transplant
  Mean calculated ALT (U/L)
Average graft function as assessed by ALT | 4 years post-transplant
  Mean calculated ALT (U/L)
Average graft function as assessed by bilirubin | 1 year post-transplant
  Mean calculated bilirubin (mg/dL)
Average graft function as assessed by bilirubin | 2 years post-transplant
  Mean calculated bilirubin (mg/dL)
Average graft function as assessed by bilirubin | 3 years post-transplant
  Mean calculated bilirubin (mg/dL)
Average graft function as assessed by Bilirubin | 4 years post-transplant
  Mean calculated bilirubin (mg/dL)
Graft function as assessed by Mean calculated Model for End Stage Liver Disease (MELD) score | 1 year post-transplant
  Mean calculated MELD score. MELD score indicates the severity of liver disease, with scores ranging from 0-40. The higher the score the more severe the disease
Graft function as assessed by Mean calculated MELD score | 2 years post-transplant
  Mean calculated MELD score. MELD score indicates the severity of liver disease, with scores ranging from 0-40. The higher the score the more severe the disease
Graft function as assessed by Mean calculated MELD score | 3 years post-transplant
  Mean calculated MELD score. MELD score indicates the severity of liver disease, with scores ranging from 0-40. The higher the score the more severe the disease
Graft function as assessed by Mean calculated MELD score | 4 years post-transplant
  Mean calculated MELD score. MELD score indicates the severity of liver disease, with scores ranging from 0-40. The higher the score the more severe the disease
Graft function as assessed by AST to Platelet Ratio (APRI) index | 1 year post-transplant
  Mean calculated APRI index [( AST / upper limits of normal (ULN) AST ) x 100] / Platelets (109/L)] An APRI score greater than 1.0 has a sensitivity of 76% and specificity of 72% for predicting cirrhosis. In addition, APRI score greater than 0.7 has a sensitivity of 77% and specificity of 72% for predicting significant hepatic fibrosis.For detection of cirrhosis, using an APRI cutoff score of 2.0 is more specific (91%) but less sensitive (46%). The lower the APRI score (less than 0.5), the greater the negative predictive value (and ability to rule out cirrhosis) and the higher the value (greater than 1.5) the greater the positive predictive value (and ability to rule in cirrhosis); midrange values are less helpful.
Graft function as assessed by AST to Platelet Ratio (APRI) index | 2 years post-transplant
  Mean calculated APRI index [( AST / ULN AST ) x 100] / Platelets (109/L)] An APRI score greater than 1.0 has a sensitivity of 76% and specificity of 72% for predicting cirrhosis. In addition, APRI score greater than 0.7 has a sensitivity of 77% and specificity of 72% for predicting significant hepatic fibrosis.For detection of cirrhosis, using an APRI cutoff score of 2.0 is more specific (91%) but less sensitive (46%). The lower the APRI score (less than 0.5), the greater the negative predictive value (and ability to rule out cirrhosis) and the higher the value (greater than 1.5) the greater the positive predictive value (and ability to rule in cirrhosis); midrange values are less helpful.
Graft function as assessed by AST to Platelet Ratio (APRI) index | 3 years post-transplant
  Mean calculated APRI index [( AST / ULN AST ) x 100] / Platelets (109/L)] An APRI score greater than 1.0 has a sensitivity of 76% and specificity of 72% for predicting cirrhosis. In addition, APRI score greater than 0.7 has a sensitivity of 77% and specificity of 72% for predicting significant hepatic fibrosis.For detection of cirrhosis, using an APRI cutoff score of 2.0 is more specific (91%) but less sensitive (46%). The lower the APRI score (less than 0.5), the greater the negative predictive value (and ability to rule out cirrhosis) and the higher the value (greater than 1.5) the greater the positive predictive value (and ability to rule in cirrhosis); midrange values are less helpful.
Graft function as assessed by AST to Platelet Ratio (APRI) index | 4 years post-transplant
  Mean calculated APRI index [( AST / ULN AST ) x 100] / Platelets (109/L)] An APRI score greater than 1.0 has a sensitivity of 76% and specificity of 72% for predicting cirrhosis. In addition, APRI score greater than 0.7 has a sensitivity of 77% and specificity of 72% for predicting significant hepatic fibrosis.For detection of cirrhosis, using an APRI cutoff score of 2.0 is more specific (91%) but less sensitive (46%). The lower the APRI score (less than 0.5), the greater the negative predictive value (and ability to rule out cirrhosis) and the higher the value (greater than 1.5) the greater the positive predictive value (and ability to rule in cirrhosis); midrange values are less helpful.
Metabolic Outcome as assessed by Body mass index (BMI) | 1 year post-transplant
  Mean calculated BMI (weight in kilograms/height in meters squared)
Metabolic Outcome as assessed by Body mass index (BMI) | 2 years post-transplant
  Mean calculated BMI(weight in kilograms/height in meters squared)
Metabolic Outcome as assessed by Body mass index (BMI) | 3 years post-transplant
  Mean calculated BMI(weight in kilograms/height in meters squared)
Metabolic Outcome as assessed by Body mass index (BMI) | 4 years post-transplant
  Mean calculated BMI(weight in kilograms/height in meters squared)
Average hemoglobin a1c among participants at 1 year | 1 years post-transplant
  Mean calculated hemoglobin a1c (mg/dL)
Average hemoglobin a1c among participants at 2 years | 2 years post-transplant
  Mean calculated hemoglobin a1c (mg/dL)
Average hemoglobin a1c among participants at 3 years | 3 years post-transplant
  Mean calculated hemoglobin a1c (mg/dL)
Average hemoglobin a1c among participants at 4 years | 4 years post-transplant
  Mean calculated hemoglobin a1c (mg/dL)
Number of HIV breakthroughs | From date of transplant through end of follow-up, up to 4 years
  Measured by local sites' Clinical Laboratory Improvement Amendments (CLIA) certified lab with episode of HIV breakthrough defined as 2 consecutive plasma HIV viral loads >200 copies/mL or one HIV viral load >1000 copies/mL after a period of virologic control post-transplant
Number of opportunistic infections | From date of transplant through end of follow-up, up to 4 years
  Cumulative incidence of opportunistic infections
Number of X4 tropic virus breakthroughs | From date of transplant through end of follow-up, up to 4 years
  Measured by sending virus at time of breakthrough for HIV co-receptor assay
Number of vascular complications | From date of transplant through year 1
  Number of vascular complications within 1 year of transplant, e.g. thrombosis, aneurysm
Number of surgical complications | From date of transplant through year 1
  Number of surgical complications within 1 year of transplant, e.g. delayed closure, wound dehiscence
Number of viral-related malignancies | From date of transplant through end of follow-up, up to 4 years
  Number of malignancies as determined by local pathology
Hepatitis C (HCV) sustained viral response post-transplant | 12 weeks HCV treatment
  Proportion of HCV RNA positive recipients that achieve a sustained virologic response week 12 post-treatment (<15 IU/mL) with direct acting antivirals
Number of the formation of de novo donor-specific human leukocyte antigen(HLA) antibodies | From date of transplant through end of year 1
  Proportion of participants with a de novo donor-specific HLA antibody as measured and reported by local sites' lab
Time to first occurrence of all-cause-mortality or graft failure or renal allograft rejection or HIV breakthrough or HIV virologic failure or AIDS defining illness as a composite measure | From date of transplant through end of follow-up, up to 4 years
  Time to first of any of these events: all-cause-mortality or graft failure or renal allograft rejection or HIV breakthrough or HIV virologic failure or AIDS defining illness

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (26):
- United States (26):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York University School of Medicine, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee Health and Science Center, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Benner SE, Zhu X, Hussain S, Florman S, Eby Y, Fernandez RE, Ostrander D, Rana M, Ottmann S, Hand J, Price JC, Pereira MR, Wojciechowski D, Simkins J, Stosor V, Mehta SA, Aslam S, Malinis M, Haidar G, Massie A, Smith ML, Odim J, Morsheimer M, Quinn TC, Laird GM, Siliciano R, Balagopal A, Segev DL, Durand CM, Redd AD, Tobian AAR. HIV-Positive Liver Transplant Does not Alter the Latent Viral Reservoir in Recipients With Antiretroviral Therapy-Suppressed HIV. J Infect Dis. 2023 Nov 2;228(9):1274-1279. doi: 10.1093/infdis/jiad241. PMID 37379584
- [Derived] Werbel WA, Brown DM, Kusemiju OT, Doby BL, Seaman SM, Redd AD, Eby Y, Fernandez RE, Desai NM, Miller J, Bismut GA, Kirby CS, Schmidt HA, Clarke WA, Seisa M, Petropoulos CJ, Quinn TC, Florman SS, Huprikar S, Rana MM, Friedman-Moraco RJ, Mehta AK, Stock PG, Price JC, Stosor V, Mehta SG, Gilbert AJ, Elias N, Morris MI, Mehta SA, Small CB, Haidar G, Malinis M, Husson JS, Pereira MR, Gupta G, Hand J, Kirchner VA, Agarwal A, Aslam S, Blumberg EA, Wolfe CR, Myer K, Wood RP, Neidlinger N, Strell S, Shuck M, Wilkins H, Wadsworth M, Motter JD, Odim J, Segev DL, Durand CM, Tobian AAR; HOPE in Action Investigators. National Landscape of Human Immunodeficiency Virus-Positive Deceased Organ Donors in the United States. Clin Infect Dis. 2022 Jun 10;74(11):2010-2019. doi: 10.1093/cid/ciab743. PMID 34453519